CLINICAL TRIAL: NCT05444387
Title: The Effect of Upper Limb Loading With External Weights During Partial Body Weight Support Treadmill Training on Gait and Trunk Control in Ambulatory Children With Cerebral Palsy: A Randomized Controlled Trial
Brief Title: The Effect of Upper Limb Loading During Partial Body Weight Support Treadmill Training in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Alya Abdelghafour Alkhajeh (Other)
Responsible Party: Sponsor-Investigator, Alya Abdelghafour Alkhajeh, Postgraduate Student, University of Sharjah
Organization: University of Sharjah (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U19102427
Record Dates: First submitted 2022-06-19; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper Limb Loading Group (Experimental): Partial body weight support treadmill training with upper limb external weights in addition to conventional treatment: balance, gait training, facilitation for normal development
  Interventions: Other: Upper limb loading
- Control Group (No Intervention): Partial body weight support treadmill training without upper limb external weights in addition to conventional treatment: balance, gait training, facilitation for normal development

INTERVENTIONS:
Other: Upper limb loading — 1 lb. external weight will be wrapped around both wrists during partial body weight support treadmill training. The partial body weight support treadmill training will be given for a maximum of 30 minutes and will finish earlier if the child asked to stop, or if the child stopped stepping. Body weight support will be systematically reduced, walking speed will be progressively increased over the training period, upright standing posture will be emphasized and normal kinematic components of the gait cycle will be facilitated during the training session. The training protocol for the current study will consist of 2 training sessions per weeks with at least one day in between and will last for 6 weeks.
  Arms: Upper Limb Loading Group

SUMMARY:
Objectives:

To look for the effect of upper limb loading with external weights during partial body weight support treadmill training on gait speed, gait endurance and trunk control.

Hypothesis:

Investigator's hypothesis is that loading the upper limb with 1 lb. external weights during partial body weight support treadmill training is more effective than partial body weight support treadmill training without loading of the upper limbs in improving gait speed, gait endurance and trunk control.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a non-progressive neurodevelopmental disorder which affects the child's motor and sensory system, and consequently posture and walking. The underlying etiology is considered multifactorial, and no specific etiological factor has been blamed. While it may be seen in the prenatal, neonatal, and postnatal period, prenatal factors account for 70 to 80 % of all cases. Although the incidence of cerebral palsy widely varies worldwide, it has been often estimated as 1.5 to 2.5/1000. While the prevalence in young people is as high as 74%. One of the characteristics of CP is gait abnormalities because of myasthenia, spasticity and impairment of movement. Children with CP have difficulties in activities, which severely affect the children's quality of life. There is no cure for CP. WHO considers limb movement function as the main rehabilitation goal. Walking capacity training of CP needs to be taken seriously. Physiotherapy is considered the core part of CP children rehabilitation due to the risk of neurosurgery and side effects of drug intervention.

Many of the gait deviations observed in neurologically impaired patient results from their inability to adequately bear weight through their affected lower extremities during the loading phase of the gait cycle. Treadmill walking with partial body weight support (PBWS) using a harness seems to address the problem. It allows even a patient with severe weakness of lower limb extensor muscles to go through the gait cycle because lower levels of muscle forces are needed to support the body mass compared with over ground walking. In addition, the harness provides a sense of secure to the patient who has fear of falling.

Partial body weight support (PBWS) systems have been widely used as an alternative therapeutic strategy for gait training in different populations, including individuals with stroke , Parkinson's disease , Spinal cord injury and children with cerebral palsy.

Some individual studies suggested that treadmill training with body weight support was superior to treadmill training alone. The addition of body weight support makes repetitive training far more feasible for a boarder range of clients and allows for more flexibility in terms of optimizing speed and training kinematic patterns for those with weakness of other impairments limiting their gait function by increasing safety and decreasing the physical work necessary by one of more therapists. Many studies showed the effectiveness of body weight support training on gait and gross motor function in the rehabilitation of CP.

The trunk plays a critical role in the organization of postural reaction. The primary contribution of the trunk muscles is to stabilize the spine and trunk, and this stabilization is essential for free and selective movements of the head and the extremities. Children with CP frequently show impaired trunk control, which can affect performance of activities of daily life such as sitting, reaching and walking. The trunk was described as a key segment in the organization of postural stabilization and orientation control.

Upper body movement during walking provide information about balance control and gait stability, and children with CP exhibit a general increase of upper body acceleration compared to typically developing (TD) children which present a progressive decrease of acceleration from pelvis to head. Also, it has been found that excessive arm swing significantly increases local dynamics stability of human gait. And children with CP appear to rely on 'guard' arm posture as a compensation strategy to maintain balance while walking compared to newly walking toddlers. Spasticity and associated movements are also important contributing factors. The hand position of children with unilateral CP has been found to be more elevated and anterior, and their upper arm was rotated more posterior than typically developing children. A study showed that facilitation of arm swing in specific situations possibly enhances safety and reduces the risk of falling in children with CP. Using arm cycling exercise has been found as an effective method for improving both arm swing and leg angular displacements during gait of children with hemiplegic CP. Also, it has been found that bilateral upper extremity exercises has a positive effect on trunk performance and alignment in stroke patients. From all of this physiotherapists get to know the importance of involving the upper limbs in the rehabilitation program for children with CP to improve gait.

A study indicated that walking while moving hand weights through large range of motion provides a combined upper and lower body aerobic stimulus that is sufficient for endurance training for persons with poor to excellent levels of aerobic fitness. Other studies looked for the physiological effect of hand-held weights during walking in normal adults. However, according to our knowledge no studies looked for the effect of upper limb external weights on gait and trunk in children with cerebral palsy. The investigators expect that placing an external weight around the both wrists while walking on the treadmill with partial body weight support will improve trunk control and gait in ambulatory children with cerebral palsy. The purpose of this study is to investigate if adding upper limb external weights during gait training using PBWS can increase the walking endurance, speed and trunk control in ambulatory children with CP.

Objectives:

To look for the effect of upper limb loading with external weights during partial body weight support treadmill training on gait speed, gait endurance and trunk control.

Hypothesis:

Investigator's hypothesis is that loading the upper limb with 1 lb. external weights during partial body weight support treadmill training is more effective than partial body weight support treadmill training without loading of the upper limbs in improving gait speed, gait endurance and trunk control.

Trial Design:

Randomized control trial

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP confirmed by the neurologist
* Age between 4 to 8 years
* Both genders
* The level of gross motor function is between level I and II according to Gross Motor Function Classification System (GMFCS)
* The degree of spasticity according to Modified Ashworth Scale range between grade 1 and grade 2
* Children should be cognitively competent with IQ level not less than 60% and able to understand and follow instructions, as well as, in general they are cooperative
* Only Arabic and English speakers will be recruited in the study

Exclusion Criteria:

* Had any orthopedic surgery or spasticity altering procedure in the previous 12 months
* Children with visual, auditory, vestibular or perceptual deficits.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline 10-meters walk test at 6 weeks | At the baseline (before treatment starts) and 6 weeks (at the end of the treatment)
  It it a measure of walking performance because it has been shown to 1- provide a useful measure of walking endurance, 2- be a representative measure of a child's community walking speed, and 3- have 95% confidence interval (CI 0.77-0.99) in children with CP. 4- valid.
Change from Baseline Trunk Control Measurement scale at 6 weeks | At the baseline (before treatment starts) and 6 weeks (at the end of the treatment)
  It measures the trunk control level as it helps in differentiating between children who are independent in self-care and mobility and those who are not, it is valid, and it has a good reliability in children with neurological disorders.
  Trunk control Measurement Scale (TCMS) is an objective outcome measure to score trunk ability in sitting. It does consists of static and dynamic sitting balance; the latter is divided into selective movement control and dynamic reaching. The maximum value is 58 and the minimum is 0. Higher values correlate to better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Hegazy, Principal Investigator — UOS
Locations (1):
- Al Qassimi Women's and Children's Hospital, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum PL, Walter SD, Hanna SE, Palisano RJ, Russell DJ, Raina P, Wood E, Bartlett DJ, Galuppi BE. Prognosis for gross motor function in cerebral palsy: creation of motor development curves. JAMA. 2002 Sep 18;288(11):1357-63. doi: 10.1001/jama.288.11.1357. PMID 12234229
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Drougia A, Giapros V, Krallis N, Theocharis P, Nikaki A, Tzoufi M, Andronikou S. Incidence and risk factors for cerebral palsy in infants with perinatal problems: a 15-year review. Early Hum Dev. 2007 Aug;83(8):541-7. doi: 10.1016/j.earlhumdev.2006.10.004. Epub 2006 Dec 26. PMID 17188824
- [Background] Ostojic K, Paget SP, Morrow AM. Management of pain in children and adolescents with cerebral palsy: a systematic review. Dev Med Child Neurol. 2019 Mar;61(3):315-321. doi: 10.1111/dmcn.14088. Epub 2018 Oct 31. PMID 30378122
- [Background] Yu Y, Chen X, Cao S, Wu D, Zhang X, Chen X. Gait synergetic neuromuscular control in children with cerebral palsy at different gross motor function classification system levels. J Neurophysiol. 2019 May 1;121(5):1680-1691. doi: 10.1152/jn.00580.2018. Epub 2019 Mar 20. PMID 30892974
- [Background] Pinto TPS, Fonseca ST, Goncalves RV, Souza TR, Vaz DV, Silva PLP, Mancini MC. Mechanisms contributing to gait speed and metabolic cost in children with unilateral cerebral palsy. Braz J Phys Ther. 2018 Jan-Feb;22(1):42-48. doi: 10.1016/j.bjpt.2017.06.015. Epub 2017 Jul 5. PMID 28728959
- [Background] Degelaen M, De Borre L, Buyl R, Kerckhofs E, De Meirleir L, Dan B. Effect of supporting 3D-garment on gait postural stability in children with bilateral spastic cerebral palsy. NeuroRehabilitation. 2016 Jun 23;39(2):175-81. doi: 10.3233/NRE-161349. PMID 27341370
- [Background] Sewell MD, Eastwood DM, Wimalasundera N. Managing common symptoms of cerebral palsy in children. BMJ. 2014 Sep 25;349:g5474. doi: 10.1136/bmj.g5474. No abstract available. PMID 25255910
- [Background] Keeratisiroj O, Thawinchai N, Siritaratiwat W, Buntragulpoontawee M, Pratoomsoot C. Prognostic predictors for ambulation in children with cerebral palsy: a systematic review and meta-analysis of observational studies. Disabil Rehabil. 2018 Jan;40(2):135-143. doi: 10.1080/09638288.2016.1250119. Epub 2016 Nov 16. PMID 27848255
- [Background] Colver A, Fairhurst C, Pharoah PO. Cerebral palsy. Lancet. 2014 Apr 5;383(9924):1240-9. doi: 10.1016/S0140-6736(13)61835-8. Epub 2013 Nov 20. PMID 24268104
- [Background] Taflampas G, Kilbride C, Levin W, Lavelle G, Ryan JM. Interventions to Improve or Maintain Lower-Limb Function Among Ambulatory Adolescents with Cerebral Palsy: A Cross-Sectional Survey of Current Practice in the UK. Phys Occup Ther Pediatr. 2018 Nov;38(4):355-369. doi: 10.1080/01942638.2017.1400490. Epub 2017 Dec 8. PMID 29220616
- [Background] Shepherd, R., & Carr, J. (1999). Treadmill Walking in Neurorehabilitation. Neurorehabilitation and Neural Repair, 13(3), 171-173. doi:10.1177/154596839901300303
- [Background] DePaul VG, Wishart LR, Richardson J, Lee TD, Thabane L. Varied overground walking-task practice versus body-weight-supported treadmill training in ambulatory adults within one year of stroke: a randomized controlled trial protocol. BMC Neurol. 2011 Oct 21;11:129. doi: 10.1186/1471-2377-11-129. PMID 22018267
- [Background] Sousa CO, Barela JA, Prado-Medeiros CL, Salvini TF, Barela AM. Gait training with partial body weight support during overground walking for individuals with chronic stroke: a pilot study. J Neuroeng Rehabil. 2011 Aug 24;8:48. doi: 10.1186/1743-0003-8-48. PMID 21864373
- [Background] Sullivan KJ, Knowlton BJ, Dobkin BH. Step training with body weight support: effect of treadmill speed and practice paradigms on poststroke locomotor recovery. Arch Phys Med Rehabil. 2002 May;83(5):683-91. doi: 10.1053/apmr.2002.32488. PMID 11994808
- [Background] Hesse S, Konrad M, Uhlenbrock D. Treadmill walking with partial body weight support versus floor walking in hemiparetic subjects. Arch Phys Med Rehabil. 1999 Apr;80(4):421-7. doi: 10.1016/s0003-9993(99)90279-4. PMID 10206604
- [Background] Gama GL, Celestino ML, Barela JA, Forrester L, Whitall J, Barela AM. Effects of Gait Training With Body Weight Support on a Treadmill Versus Overground in Individuals With Stroke. Arch Phys Med Rehabil. 2017 Apr;98(4):738-745. doi: 10.1016/j.apmr.2016.11.022. Epub 2016 Dec 27. PMID 28034719
- [Background] Ganesan M, Sathyaprabha TN, Pal PK, Gupta A. Partial Body Weight-Supported Treadmill Training in Patients With Parkinson Disease: Impact on Gait and Clinical Manifestation. Arch Phys Med Rehabil. 2015 Sep;96(9):1557-65. doi: 10.1016/j.apmr.2015.05.007. Epub 2015 May 23. PMID 26008873
- [Background] Ganesan M, Sathyaprabha TN, Gupta A, Pal PK. Effect of partial weight-supported treadmill gait training on balance in patients with Parkinson disease. PM R. 2014 Jan;6(1):22-33. doi: 10.1016/j.pmrj.2013.08.604. Epub 2013 Sep 8. PMID 24021298
- [Background] Terson de Paleville D, McKay W, Aslan S, Folz R, Sayenko D, Ovechkin A. Locomotor step training with body weight support improves respiratory motor function in individuals with chronic spinal cord injury. Respir Physiol Neurobiol. 2013 Dec 1;189(3):491-7. doi: 10.1016/j.resp.2013.08.018. Epub 2013 Aug 31. PMID 23999001
- [Background] Willoughby KL, Dodd KJ, Shields N, Foley S. Efficacy of partial body weight-supported treadmill training compared with overground walking practice for children with cerebral palsy: a randomized controlled trial. Arch Phys Med Rehabil. 2010 Mar;91(3):333-9. doi: 10.1016/j.apmr.2009.10.029. PMID 20298820
- [Background] Mattern-Baxter K. Effects of partial body weight supported treadmill training on children with cerebral palsy. Pediatr Phys Ther. 2009 Spring;21(1):12-22. doi: 10.1097/PEP.0b013e318196ef42. PMID 19214072
- [Background] Cherng RJ, Liu CF, Lau TW, Hong RB. Effect of treadmill training with body weight support on gait and gross motor function in children with spastic cerebral palsy. Am J Phys Med Rehabil. 2007 Jul;86(7):548-55. doi: 10.1097/PHM.0b013e31806dc302. PMID 17581289
- [Background] Damiano DL, DeJong SL. A systematic review of the effectiveness of treadmill training and body weight support in pediatric rehabilitation. J Neurol Phys Ther. 2009 Mar;33(1):27-44. doi: 10.1097/NPT.0b013e31819800e2. PMID 19265768
- [Background] Aras B, Yasar E, Kesikburun S, Turker D, Tok F, Yilmaz B. Comparison of the effectiveness of partial body weight-supported treadmill exercises, robotic-assisted treadmill exercises, and anti-gravity treadmill exercises in spastic cerebral palsy. Turk J Phys Med Rehabil. 2019 Nov 22;65(4):361-370. doi: 10.5606/tftrd.2019.3078. eCollection 2019 Jun. PMID 31893273
- [Background] Flores MB, Da Silva CP. Trunk control and gross motor outcomes after body weight supported treadmill training in young children with severe cerebral palsy: a non-experimental case series. Dev Neurorehabil. 2019 Oct;22(7):499-503. doi: 10.1080/17518423.2018.1527862. Epub 2018 Oct 5. PMID 30289316
- [Background] Sharan D, Rajkumar JS, Balakrishnan R, Kulkarni A, Selvakumar K, Gampa S, Mohandoss M, Ranganathan R. Effectiveness of a low-cost body weight support training device in the rehabilitation of cerebral palsy. J Rehabil Assist Technol Eng. 2016 Nov 29;3:2055668316676047. doi: 10.1177/2055668316676047. eCollection 2016 Jan-Dec. PMID 31186916
- [Background] Su IY, Chung KK, Chow DH. Treadmill training with partial body weight support compared with conventional gait training for low-functioning children and adolescents with nonspastic cerebral palsy: a two-period crossover study. Prosthet Orthot Int. 2013 Dec;37(6):445-53. doi: 10.1177/0309364613476532. Epub 2013 Feb 22. PMID 23436693
- [Background] Dodd KJ, Foley S. Partial body-weight-supported treadmill training can improve walking in children with cerebral palsy: a clinical controlled trial. Dev Med Child Neurol. 2007 Feb;49(2):101-5. doi: 10.1111/j.1469-8749.2007.00101.x. PMID 17253995
- [Background] Verheyden G, Nieuwboer A, Mertin J, Preger R, Kiekens C, De Weerdt W. The Trunk Impairment Scale: a new tool to measure motor impairment of the trunk after stroke. Clin Rehabil. 2004 May;18(3):326-34. doi: 10.1191/0269215504cr733oa. PMID 15137564
- [Background] Bertenthal B, Von Hofsten C. Eye, head and trunk control: the foundation for manual development. Neurosci Biobehav Rev. 1998 Jul;22(4):515-20. doi: 10.1016/s0149-7634(97)00038-9. PMID 9595563
- [Background] Saavedra S, Karve SJ, Woollacott M, van Donkelaar P. Eye hand coordination in children with cerebral palsy. Exp Brain Res. 2009 Jan;192(2):155-65. doi: 10.1007/s00221-008-1549-8. Epub 2008 Oct 2. PMID 18830589
- [Background] Saavedra S, Woollacott M, van Donkelaar P. Head stability during quiet sitting in children with cerebral palsy: effect of vision and trunk support. Exp Brain Res. 2010 Feb;201(1):13-23. doi: 10.1007/s00221-009-2001-4. Epub 2009 Sep 16. PMID 19756550
- [Background] Verheyden G, Vereeck L, Truijen S, Troch M, Herregodts I, Lafosse C, Nieuwboer A, De Weerdt W. Trunk performance after stroke and the relationship with balance, gait and functional ability. Clin Rehabil. 2006 May;20(5):451-8. doi: 10.1191/0269215505cr955oa. PMID 16774097
- [Background] Verheyden G, Nieuwboer A, De Wit L, Feys H, Schuback B, Baert I, Jenni W, Schupp W, Thijs V, De Weerdt W. Trunk performance after stroke: an eye catching predictor of functional outcome. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):694-8. doi: 10.1136/jnnp.2006.101642. Epub 2006 Dec 18. PMID 17178824
- [Background] Hadders-Algra M & Brogren E. Postural control: A key issue in developmental disorders (1st ed.). London: MacKeith Press; 2008.
- [Background] Prosser LA, Lee SC, VanSant AF, Barbe MF, Lauer RT. Trunk and hip muscle activation patterns are different during walking in young children with and without cerebral palsy. Phys Ther. 2010 Jul;90(7):986-97. doi: 10.2522/ptj.20090161. Epub 2010 Apr 29. PMID 20430948
- [Background] van der Heide JC, Fock JM, Otten B, Stremmelaar E, Hadders-Algra M. Kinematic characteristics of postural control during reaching in preterm children with cerebral palsy. Pediatr Res. 2005 Sep;58(3):586-93. doi: 10.1203/01.pdr.0000176834.47305.26. PMID 16148078
- [Background] Assaiante C, Mallau S, Viel S, Jover M, Schmitz C. Development of postural control in healthy children: a functional approach. Neural Plast. 2005;12(2-3):109-18; discussion 263-72. doi: 10.1155/NP.2005.109. PMID 16097479
- [Background] Summa A, Vannozzi G, Bergamini E, Iosa M, Morelli D, Cappozzo A. Multilevel Upper Body Movement Control during Gait in Children with Cerebral Palsy. PLoS One. 2016 Mar 21;11(3):e0151792. doi: 10.1371/journal.pone.0151792. eCollection 2016. PMID 26999362
- [Background] Punt M, Bruijn SM, Wittink H, van Dieen JH. Effect of arm swing strategy on local dynamic stability of human gait. Gait Posture. 2015 Feb;41(2):504-9. doi: 10.1016/j.gaitpost.2014.12.002. Epub 2014 Dec 26. PMID 25582804
- [Background] Meyns P, Desloovere K, Van Gestel L, Massaad F, Smits-Engelsman B, Duysens J. Altered arm posture in children with cerebral palsy is related to instability during walking. Eur J Paediatr Neurol. 2012 Sep;16(5):528-35. doi: 10.1016/j.ejpn.2012.01.011. Epub 2012 Feb 14. PMID 22336190
- [Background] Delabastita T, Desloovere K, Meyns P. Restricted Arm Swing Affects Gait Stability and Increased Walking Speed Alters Trunk Movements in Children with Cerebral Palsy. Front Hum Neurosci. 2016 Jul 15;10:354. doi: 10.3389/fnhum.2016.00354. eCollection 2016. PMID 27471457
- [Background] Hussein, Z. A., Abd-Elwahab, M. S., & El-Shennawy, S. A. (2014). Effect of arm cycling on gait of children with hemiplegic cerebral palsy. Egyptian Journal of Medical Human Genetics, 15(3), 273-279. doi:10.1016/j.ejmhg.2014.02.008
- [Background] Lee DH, Park SH, Han JW. Effect of bilateral upper extremity exercise on trunk performance in patients with stroke. J Phys Ther Sci. 2017 Apr;29(4):625-628. doi: 10.1589/jpts.29.625. Epub 2017 Apr 20. PMID 28533598
- [Background] Awad A, Shaker H, Shendy W, Fahmy M. Effect of shoulder girdle strengthening on trunk alignment in patients with stroke. J Phys Ther Sci. 2015 Jul;27(7):2195-200. doi: 10.1589/jpts.27.2195. Epub 2015 Jul 22. PMID 26311953
- [Background] Auble TE, Schwartz L, Robertson RJ. Aerobic Requirements for Moving Handweights Through Various Ranges of Motion While Walking. Phys Sportsmed. 1987 Jun;15(6):133-40. doi: 10.1080/00913847.1987.11709378. PMID 27404531
- [Background] Owens SG, al-Ahmed A, Moffatt RJ. Physiological effects of walking and running with hand-held weights. J Sports Med Phys Fitness. 1989 Dec;29(4):384-7. PMID 2628637
- [Background] Graves JE, Pollock ML, Montain SJ, Jackson AS, O'Keefe JM. The effect of hand-held weights on the physiological responses to walking exercise. Med Sci Sports Exerc. 1987 Jun;19(3):260-5. PMID 3600240
- [Background] Swe NN, Sendhilnnathan S, van Den Berg M, Barr C. Over ground walking and body weight supported walking improve mobility equally in cerebral palsy: a randomised controlled trial. Clin Rehabil. 2015 Nov;29(11):1108-16. doi: 10.1177/0269215514566249. Epub 2015 Jan 30. PMID 25636992
- [Background] Fedrizzi E, Facchin P, Marzaroli M, Pagliano E, Botteon G, Percivalle L, Fazzi E. Predictors of independent walking in children with spastic diplegia. J Child Neurol. 2000 Apr;15(4):228-34. doi: 10.1177/088307380001500405. PMID 10805188
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Elbasatiny, H., & Abdelaziem, A. (2015). Effect of Trunk Exercises on Trunk control, Balance and Mobility Function in Children with Hemiparetic Cerebral Palsy. International Journal of Therapies and Rehabilitation Research, 4(5), 236. doi:10.5455/ijtrr.00000094
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Demura, S., Yamaji, S., Kitabayashi, T., Yamada, T., & Uchiyama, M. (2007). Effects of the package holding with one hand on the center of foot pressure. Sport Sciences for Health, 2(2), 58-63. doi:10.1007/s11332-007-0040-4
- [Background] Ibrahim AI, Alhusaini AA, Hegazy FA, Hawamdeh ZM. Effectiveness of foot wedge and carrying weighted bag on loading the paretic lower limb in children with hemiparetic cerebral palsy. NeuroRehabilitation. 2013;32(3):563-71. doi: 10.3233/NRE-130878. PMID 23648610
- [Background] Meyer-Heim A, Borggraefe I, Ammann-Reiffer C, Berweck S, Sennhauser FH, Colombo G, Knecht B, Heinen F. Feasibility of robotic-assisted locomotor training in children with central gait impairment. Dev Med Child Neurol. 2007 Dec;49(12):900-6. doi: 10.1111/j.1469-8749.2007.00900.x. PMID 18039236
- [Background] Pirpiris M, Wilkinson AJ, Rodda J, Nguyen TC, Baker RJ, Nattrass GR, Graham HK. Walking speed in children and young adults with neuromuscular disease: comparison between two assessment methods. J Pediatr Orthop. 2003 May-Jun;23(3):302-7. PMID 12724591
- [Background] Chrysagis N, Skordilis EK, Koutsouki D. Validity and clinical utility of functional assessments in children with cerebral palsy. Arch Phys Med Rehabil. 2014 Feb;95(2):369-74. doi: 10.1016/j.apmr.2013.10.025. Epub 2013 Nov 12. PMID 24239880
- [Background] Pham HP, Eidem A, Hansen G, Nyquist A, Vik T, Saether R. Validity and Responsiveness of the Trunk Impairment Scale and Trunk Control Measurement Scale in Young Individuals with Cerebral Palsy. Phys Occup Ther Pediatr. 2016 Nov;36(4):440-52. doi: 10.3109/01942638.2015.1127867. Epub 2016 Feb 18. PMID 26890372
- [Background] Marsico P, Mitteregger E, Balzer J, van Hedel HJA. The Trunk Control Measurement Scale: reliability and discriminative validity in children and young people with neuromotor disorders. Dev Med Child Neurol. 2017 Jul;59(7):706-712. doi: 10.1111/dmcn.13425. Epub 2017 Apr 4. PMID 28374541
- [Derived] Alkhajeh A, Arumugam A, Abd ElKafy E, Hegazy F. The effect of upper limb loading with external weights on gait and trunk control in ambulatory children with spastic hemiplegic cerebral palsy: a randomized controlled trial. Eur Rev Med Pharmacol Sci. 2024 Mar;28(6):2117-2126. doi: 10.26355/eurrev_202403_35715. PMID 38567574